CLINICAL TRIAL: NCT07199387
Title: PeerOnCall: A Cluster Randomized Trial of a Peer Support Mobile Health Platform in Canadian Fire Service Organizations
Brief Title: PeerOnCall: Implementing and Evaluating App-Based Peer Support in Canadian Fire Services
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Sandra Moll, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 204097; 204097 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Firefighters
Keywords: Peer Support; Mobile Health Applications; Mental Health; Firefighters; Occupational Health; Workplace Wellbeing; Implementation Science
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App Users (Structured Implementation) (Experimental): All participating organizations will receive access to PeerOnCall, a mobile mental health and peer support platform co-designed by and for Canadian public safety providers (PSP) that includes: a) an app for frontline workers, b) an app for peer support providers, and c) an administrative portal for organizational leaders. The structured implementation (intervention) group will follow a structured protocol designed to promote weekly app engagement.
  Interventions: Other: App Users (Structured Implementation)
- App Users (Standard Implementation) (Active Comparator): All participating organizations will receive access to PeerOnCall, a mobile mental health and peer support platform co-designed by and for Canadian public safety providers (PSP) that includes: a) an app for frontline workers, b) an app for peer support providers, and c) an administrative portal for organizational leaders. The standard implementation (control) group will receive baseline support, allowing firefighters to use the app as they choose.
  Interventions: Other: App Users (Standard Implementation)

INTERVENTIONS:
Other: App Users (Structured Implementation) — The structured implementation (intervention) group will follow a structured protocol designed to promote weekly app engagement. This includes regular updates to customized content, reminders to use the app, and feedback on use. Weekly content updates and push notifications will be provided through the app, and the research team will communicate monthly with organizational champions with feedback reports on app utilization to reinforce engagement.
  Arms: App Users (Structured Implementation)
Other: App Users (Standard Implementation) — The standard implementation (control) group will receive baseline support, allowing firefighters to use the app as they choose. The research team will provide an initial orientation for organizations and peer supporters, but the organizational champion will be responsible for communication and follow-up. The research team will respond to questions and prompt data collection.
  Arms: App Users (Standard Implementation)

SUMMARY:
The goal of this clinical trial is to test how best to implement a mobile peer support app called PeerOnCall in Canadian fire services. The main questions it aims to answer are:

1. Do firefighters use the app more with a structured implementation compared to standard implementation?
2. Does using the app improve mental health and workplace outcomes? Researchers will compare a standard implementation approach with basic onboarding to more structured implementation with weekly reminders, new content, and feedback reports to see if these features encourage more consistent app use.

Participants will:

1. Use the PeerOnCall app to access private peer support and wellness resources.
2. Participate in surveys, interviews, and focus groups about their app experience and workplace environment.

ELIGIBILITY:
Inclusion Criteria:

* Must be a working aged adult (18-70)
* Must be employed in a participating Canadian Fire Service organization
* Agree to download the PeerOnCall app to their mobile phone (iPhone or Android)

Exclusion Criteria:

- Not able to access app on their smart device

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Score on the Mental Health Continuum at 1 year | From Baseline to the end of implementation at 1-year
  Impact on mental health (primary) outcome - A 10-point visual analogue scale (VAS) will be used to measure mental health status as a continuous variable, aligning with the mental health continuum commonly used in the public safety community. The scale uses color coding from 0 (green/well) to 10 (red/crisis) with strong concurrent validity (r = .60 to .74) compared to other anxiety measures. Pilot research indicated that firefighters are resistant to lengthy psychological questionnaires, so this brief, intuitive, and widely accepted single-item scale was selected to optimize response rates. App users will receive monthly in-app notifications prompting them to complete the scale. Since the scale is integrated into the app, data can be directly linked to app utilization.
App Engagement (App Opens) | From enrolment to the end of implementation at 1-year
  App opens will be tracked as a binary variable, measuring whether an employee opens the app at least once during the 12-month study period. This initial adoption measure will be monitored using unique ID numbers to track the total number of app opens per user. A list of eligible employees will be established at the start of the intervention and monitored over time to assess engagement across the organization.
App Engagement (Peer Support Outreach) | From enrolment to the end of implementation at 1-year
  Peer support outreach will be measured by the number of text or phone interactions initiated with a peer support provider. Software analytics will track individual use patterns, including whether users reach out once or multiple times to peer support. Higher outreach frequency reflects greater engagement with the app.

SECONDARY OUTCOMES:
Change from Baseline Score on the WLQ-F at 1 year | From Baseline to the end of implementation at 1-year
  The secondary outcome is firefighter work performance, measured using the 36-item Work Limitations Questionnaire for Firefighters (WLQ-F), which assesses physical, cognitive, social, emotional, and time-related work demands. Responses are scored on a 5-point Likert scale from 0% (not limited at all) to 100% (unable to do), with higher scores indicating greater limitations.
Mental Health Absenteeism | From enrolment to the end of implementation at 1-year
  Absenteeism, measured as the number of mental health related sick days will also be tracked in each organization. These productivity or performance measures provide important organizational impact data.

CONTACTS AND LOCATIONS:
Locations (1):
- 20 Fire Service Organizations across Canada, Hamilton, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moll SE, Patten S, Stuart H, MacDermid JC, Kirsh B. Beyond Silence: A Randomized, Parallel-Group Trial Exploring the Impact of Workplace Mental Health Literacy Training with Healthcare Employees. Can J Psychiatry. 2018 Dec;63(12):826-833. doi: 10.1177/0706743718766051. Epub 2018 Apr 19. PMID 29673271
- [Background] Lesage FX, Berjot S, Deschamps F. Clinical stress assessment using a visual analogue scale. Occup Med (Lond). 2012 Dec;62(8):600-5. doi: 10.1093/occmed/kqs140. Epub 2012 Sep 10. PMID 22965867
- [Background] Dutheil F, Palgen C, Brousse G, Cornet T, Mermillod M, Lakbar I, Vallet G, Baker JS, Schmidt J, Charbotel B, Pereira B, Delamarre L. Validation of visual analog scales of mood and anxiety at the workplace. PLoS One. 2024 Dec 31;19(12):e0316159. doi: 10.1371/journal.pone.0316159. eCollection 2024. PMID 39739967
- [Background] Moll SE, Ricciardelli R, Carleton RN, MacDermid JC, Czarnuch S, MacPhee RS. PeerOnCall: Evaluating Implementation of App-Based Peer Support in Canadian Public Safety Organizations. Int J Environ Res Public Health. 2025 Aug 13;22(8):1269. doi: 10.3390/ijerph22081269. PMID 40869854
- [Background] Raggi A, Bernard RM, Toppo C, Sabariego C, Salvador Carulla L, Lukersmith S, Hakkaart-van Roijen L, Merecz-Kot D, Olaya B, Antunes Lima R, Gutierrez-Marin D, Vorstenbosch E, Curatoli C, Cacciatore M. The EMPOWER Occupational e-Mental Health Intervention Implementation Checklist to Foster e-Mental Health Interventions in the Workplace: Development Study. J Med Internet Res. 2024 Mar 15;26:e48504. doi: 10.2196/48504. PMID 38488846
- [Background] Goraya NK, Alvarez E, Young M, Moll S. PeerOnCall: Exploring how organizational culture shapes implementation of a peer support app for public safety personnel. Compr Psychiatry. 2024 Nov;135:152524. doi: 10.1016/j.comppsych.2024.152524. Epub 2024 Aug 12. PMID 39146608
- [Background] Damschroder LJ, Reardon CM, Widerquist MAO, Lowery J. The updated Consolidated Framework for Implementation Research based on user feedback. Implement Sci. 2022 Oct 29;17(1):75. doi: 10.1186/s13012-022-01245-0. PMID 36309746
- [Background] Howarth A, Quesada J, Silva J, Judycki S, Mills PR. The impact of digital health interventions on health-related outcomes in the workplace: A systematic review. Digit Health. 2018 May 10;4:2055207618770861. doi: 10.1177/2055207618770861. eCollection 2018 Jan-Dec. PMID 29942631
- [Background] Voth M, Chisholm S, Sollid H, Jones C, Smith-MacDonald L, Bremault-Phillips S. Correction: Efficacy, Effectiveness, and Quality of Resilience-Building Mobile Health Apps for Military, Veteran, and Public Safety Personnel Populations: Scoping Literature Review and App Evaluation. JMIR Mhealth Uhealth. 2023 Aug 28;11:e51609. doi: 10.2196/51609. PMID 37639713
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Johnson, C. C., Vega, L., Kohalmi, A. L., Roth, J. C., Howell, B. R., & Van Hasselt, V. B. (2020). Enhancing mental health treatment for the firefighter population: Understanding fire culture, treatment barriers, practice implications, and research directions. Professional Psychology: Research and Practice, 51(3), 304-311. https://doi.org/10.1037/pro0000266
- [Background] Canadian Association of Fire Chiefs (Nov 2024). The State of Fire and Emergency services in Canada: Results of the great Canadian Fire census 2024. Ottawa: CAFC
- [Background] Carleton, R. N., Afifi, T. O., Turner, S., Taillieu, T., LeBouthillier, D. M., Duranceau, S., Sareen, J., Ricciardelli, R., MacPhee, R. S., Groll, D., Hozempa, K., Brunet, A., Weekes, J. R., Griffiths, C. T., Abrams, K. J., Jones, N. A., Beshai, S., Cramm, H. A., Dobson, K. S., . . . Asmundson, G. J. G. (2018). Suicidal ideation, plans, and attempts among public safety personnel in Canada.Canadian Psychology / Psychologie canadienne, 59(3), 220-231. https://doi.org/10.1037/cap0000136
- [Background] MacDermid JC, Lomotan M, Hu MA. Canadian Career Firefighters' Mental Health Impacts and Priorities. Int J Environ Res Public Health. 2021 Dec 1;18(23):12666. doi: 10.3390/ijerph182312666. PMID 34886394
- [Background] Carleton RN, Afifi TO, Turner S, Taillieu T, Duranceau S, LeBouthillier DM, Sareen J, Ricciardelli R, MacPhee RS, Groll D, Hozempa K, Brunet A, Weekes JR, Griffiths CT, Abrams KJ, Jones NA, Beshai S, Cramm HA, Dobson KS, Hatcher S, Keane TM, Stewart SH, Asmundson GJG. Mental Disorder Symptoms among Public Safety Personnel in Canada. Can J Psychiatry. 2018 Jan;63(1):54-64. doi: 10.1177/0706743717723825. Epub 2017 Aug 28. PMID 28845686
- See also: PeerOnCall Research Website — https://www.oncallapp.ca/research/national-research-team/